CLINICAL TRIAL: NCT05398952
Title: Post-COVID-19 Outpatient Care and Biomarkers for Persisting Symptoms of Post-COVID-19 Disease - A Prospective Registry and Biobank
Brief Title: Post-COVID-19 Outpatient Care and Biomarkers
Acronym: POSTCOV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mariann Gyongyosi, Principal Investigator, Medical University of Vienna
Other Study IDs: Protocol Version 2
Record Dates: First submitted 2022-05-31; First posted 2022-06-01 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Post Viral Fatigue; Viral Myocarditis; POTS
Keywords: long/post-COVID; multiorgan disease; biomarkers; cardiovascular imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Frozen serum and plasma samples, as well as blood samples stored in RNA and cDNA tubes; peripheral blood mononuclear cells will be separated by Ficoll and frozen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Long-COVID: Patients with previous COVID-19 disease, and having long COVID symptoms 3 months after the active infection.
  Interventions: Diagnostic Test: Laboratory investigations
- Post-COVID-19 without long-COVID syndrome: Patients with previous COVID-19 disease, without long COVID symptoms
  Interventions: Diagnostic Test: Laboratory investigations
- IcMP (positive control): Patients with ischemic heart disease without COVID-19 disease, and vaccinated at least with one injection
  Interventions: Diagnostic Test: Laboratory investigations
- Healthy (negative control): Healthy individuals without COVID-19 disease, and vaccinated at least with one injection
  Interventions: Diagnostic Test: Laboratory investigations

INTERVENTIONS:
Diagnostic Test: Laboratory investigations — Laboratory investigations correlated with symptoms and imaging results

SUMMARY:
The aims of this case-control, non-randomized study including patients with post-COVID-19 persisting symptoms are 1) to establish the large blood biobank, 2) to examine levels of circulating inflammatory biomarkers and different classes of non-coding RNAs (ncRNA), such as selected circRNAs and miRNAs, in plasma and serum samples collected from patients with post- COVID-19, 3) to test the levels of cfDNA in plasma and serum, 4) to define correlation between ncRNAs and cf-DNA with persistent clinical symptoms, and type of symptoms, and 5) to investigate diagnostic and prognostic performances of these circulating biomarkers.

Study design. This is a prospective registry including biobank.

DETAILED DESCRIPTION:
Currently, several studies are ongoing to investigate different treatment modalities of post-COVID-19 symptoms, but there is a complete lack of investigations on biomarkers predicting type, duration or severity of post-COVID-19 symptoms. The aim of this study is to investigate circulatory biomarkers diagnostic or predictive for long/post-COVID-19 syndrome.

Study patients. Patients with at least 3 weeks after proven infection by SARS-CoV-2, reflected by at least one positive PCR-test in nose throat swabs, who visits at the Post-COVID-19 outpatient clinic of the Medical University of Vienna, will be consequently recruited into the presented registry. Additionally, 100 vaccinated patients with HFrEF and 100 healthy vaccinated volunteers will be recruited to serve as comparison groups.

Methods. Identity of the registry patients will be protected by pseudonymization. During the ambulatory visit, basic clinical examination, electrocardiogram, chest X-ray, routine laboratory tests will be performed. Additionally, venous blood will be collected for biobank.

Expected Outcome This registry will provide further insights regarding pathophysiology, risk stratification and treatment of complex post-COVID-19 symptoms. Specific therapies and search of prognostic factors will enable to select patients with high risk of persistence or worsening of their symptoms thereby improve patient care.

ELIGIBILITY:
Inclusion Criteria:

For post-COVID patient group:

* Age≥18to90years
* Proven infection by SARS-CoV2, at least 3 weeks after recovery from the infection
* Signed informed consent For HFrEF patient group:

For vaccinated healthy volunteer control group:

* Full vaccination against SARS-CoV2 at least 3 weeks before inclusion in the study
* Signed informed consent

Exclusion Criteria:

* non-willingness to participate or withdrawal of informed consent
* Clinically confirmed HFrEF (EF <40%)
* participation in any SARS-CoV-2 medical treatment trial
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient clinical patients with at least 6 weeks after proven infection by SARS-CoV-2, reflected by at least one positive PCR-test in nose throat swabs, who visits at the Post-COVID-19 outpatient clinic of the Medical University of Vienna, will be consequently recruited into the presented study. A written informed consent will be present before inclusion. 100 vaccinated HFrEF patient volunteers will be recruited during routine visits to our outpatient clinic. 100 healthy, vaccinated volunteers will be recruited from among hospital staff.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in circulating biomarkers | 3 years
  circularRNA

SECONDARY OUTCOMES:
Change in circulating proteins | 3 years
  Proteomics
Change in neutralizing antibodies | 3 years
  neutralizing antibodies
Changes in ECGs | 3 years
  ECG signs
Cardiac magnetic resonance imaging abnormalities | 3 years
  Pericardial effusion

CONTACTS AND LOCATIONS:
Overall Officials: Mariann Gyöngyösi, MD PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Cardiology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request; after signature of the Data Sharing Agreement
Supporting Information: Study Protocol, ICF
Time Frame: After the study closure, and publication of the data
Access Criteria: Upon reasonable request; after signature of the Data Sharing Agreement

REFERENCES:
- [Derived] Gyongyosi M, Hasimbegovic E, Han E, Zlabinger K, Spannbauer A, Riesenhuber M, Hamzaraj K, Bergler-Klein J, Hengstenberg C, Kammerlander A, Kastl S, Loewe C, Beitzke D. Improvement of Symptoms and Cardiac Magnetic Resonance Abnormalities in Patients with Post-Acute Sequelae of SARS-CoV-2 Cardiovascular Syndrome (PASC-CVS) after Guideline-Oriented Therapy. Biomedicines. 2023 Dec 14;11(12):3312. doi: 10.3390/biomedicines11123312. PMID 38137533
- [Derived] Gyongyosi M, Lukovic D, Mester-Tonczar J, Zlabinger K, Einzinger P, Spannbauer A, Schweiger V, Schefberger K, Samaha E, Bergler-Klein J, Riesenhuber M, Nitsche C, Hengstenberg C, Mucher P, Haslacher H, Breuer M, Strassl R, Puchhammer-Stockl E, Loewe C, Beitzke D, Hasimbegovic E, Zelniker TA. Effect of monovalent COVID-19 vaccines on viral interference between SARS-CoV-2 and several DNA viruses in patients with long-COVID syndrome. NPJ Vaccines. 2023 Sep 29;8(1):145. doi: 10.1038/s41541-023-00739-2. PMID 37773184